CLINICAL TRIAL: NCT05203991
Title: Explorative Study on Occult Avascular Osteonecrosis in a Pediatric Patients Cohort With Sickle Cell Disease
Brief Title: Avascular Bone Necrosis in Sickle Cell Disease: a Pediatric Study.
Acronym: OsteoSCD
Status: Completed | Type: Observational
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Vincenzo Voi, MD, San Luigi Gonzaga Hospital
Other Study IDs: Osteonecrosis SCD
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Sickle Cell Disease
Keywords: Avascular necrosis
MeSH Terms: conditions — Anemia, Sickle Cell; Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Avascular necrosis (AVN) is a serious complication of sickle cell disease, especially in pediatric patients where the prevalence is between 3% and 8% and are more frequent in patients with multiple vaso-occlusive crisis (VOC). The prevalence of AVN is usually made by a study of the hip through radiography, whereas other possible sites of ischemic infarcts are evaluated only in case of specific symptoms. In addition, bone infarcts may be the trigger for additional VOC.

In this study, we want to investigate the presence of possible bone lesions even in asymptomatic or paucisymptomatic children.

This is a prospective interventional and monocentric study whose objective is to describe the prevalence of osteonecrosis in children with sickle cell disease in Italy

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients diagnosed with sickle cell anemia (HbSS, HbS/β0, HbS/β+, HbSC) with or without known avascular lesions
* Age ≥ 7 and < 18 years at the moment of signed consent
* Written informed consent/assent, according to local guidelines, signed by patient and/or guidelines, signed by the patient and/or at least one parent or legal guardian

Exclusion Criteria:

* - Any contraindication to perform Nuclear Magnetic Resonance Magnetic Resonance Imaging (MRI)
* Inability to obtain informed consent/assent

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sickle cell pediatric patients followed in consultation in Microcitemie Centre within the framework of their sickle cell disease at San Luigi Gonzaga Hospital, Orbassano (Turin), Italy
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Calculate the prevalence of unknown osteonecrosis | Day 1
  Avascular necrosis of the bones are diagnosed by systematic MRI at sites: total spine, femurs, shoulders, humeri and total hip. These data will be collected in the patient's medical record in patients with sickle cell anemia regardless of the number and intensity of vaso-occlusive crisis

CONTACTS AND LOCATIONS:
Locations (1):
- AOU San Luigi Gonzaga, Orbassano, Torino, Italy